CLINICAL TRIAL: NCT03539302
Title: A Prospective Randomized Multicenter Study of Flecainide Acetate Oral Inhalation Solution in Single and Repeat Dose Regimens for Acute Conversion to Sinus Rhythm in Subjects With Recent Onset of Symptomatic Paroxysmal Atrial Fibrillation
Brief Title: INhalation of Flecainide to Convert Recent Onset SympTomatic Atrial Fibrillation to siNus rhyThm (INSTANT)
Acronym: INSTANT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InCarda Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FLE-002
Record Dates: First submitted 2018-02-26; First posted 2018-05-29 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-02

CONDITIONS: Paroxysmal Atrial Fibrillation (PAF)
Keywords: Inhaled Flecainide
MeSH Terms: conditions — Atrial Fibrillation | interventions — Flecainide

STUDY DESIGN:
Intervention Model Description: The 3 parts of the study were performed sequentially. Only Part A was randomized to assign subjects to either the 30 mg dose or 60 mg. Parts B and C were not randomized. There were no comparators in this study and no masking.
Masking Description: Part A was open-label however subjects were randomized to either a single dose or a double dose. There was no masking and this was a single-arm study.
  Part B was an open-label, multicenter design to confirm the safety (including tolerability) and efficacy of the optimal dose from Part A.
  Part C was an open-label, multicenter design study to assess the feasibility of self-administration of FlecIH-103 under medical supervision. Part C also included a sub-study to evaluate a hand-held echocardiogram device to assess the feasibility of its use in an emergent setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Repeat dose inhaled flecainide acetate (Experimental): One 120 mg dose of flecainide acetate inhalation solution will be administered via two oral inhalations of 3.5 minutes. There will be a 1 minute break between the two inhalations. A single nebulizer will be used.
  A subset of enrolled patients will be included in a sub-study in which a Hand Held ECHO device at bedside will be used to confirm eligibility by verifying absence of structural heart disease. Once eligibility is confirmed the treatment for this subset of patients will be the same as described above; one 120 mg dose of flecainide acetate inhalation solution will be administered via two oral inhalations of 3.5 minutes. There will be a 1 minute break between the two inhalations. A single nebulizer will be used.
  Interventions: Drug: Flecainide Acetate

INTERVENTIONS:
Drug: Flecainide Acetate — Oral inhalation form using a nebulizer
  Other Names: FlecIH

SUMMARY:
The study consisted of 3 parts (Part A, Part B and Part C). Part A was an open-label, randomized, multi center design to evaluate the feasibility of administration of inhaled flecainide in two dosing regimens. Part B was an open-label, multicenter design to confirm the safety (including tolerability) and efficacy of the optimal inhaled flecainide dose determined from Part A. Part C was an open-label, multi center study with exploratory objectives to explore the feasibility of patient-led self administration of flecainide. Part C also included an exploratory sub-study to assess the feasibility of implementing a portable cardiac ultrasound (HHE) at screening in an emergent setting.

DETAILED DESCRIPTION:
Subjects eligible to participate in the study must provide written informed consent (IC) before randomization or any study- specific procedures.

The study consists of 3 parts (Part A, Part B and Part C) as described below:

Part A: was completed in March 2020 and was an open-label, randomized, multicenter design to evaluate the feasibility of administration of inhaled flecainide in two dosing regimens.

Subjects were randomized at a 1:1 ratio to a single (N = 10) or repeat (N = 10) dose regimen. Randomization, for the initial 20 patients in Part A was stratified by duration of the presenting AF episode (≥ 1 h up to ≤ 24 hours; > 24h up to ≤ 48h).

After completion of the 60 mg dose cohort and review of safety/tolerability and PK data, additional subjects were enrolled in an additional repeat dose regimen (90 mg estimated total lung dose (TLD), N= up to 30 subjects. An additional dose cohort of 120 mg was added to Part A which utilized a different concentration of flecainide (75 mg/mL) and formulation (FlecIH-103). The final dose of 120 mg was selected as the dose to continue evaluating in Part B.

Part B: was an open-label, multicenter design to confirm the safety (including tolerability) and efficacy of the optimal inhaled flecainide dose determined from Part A (120 mg, using the FlecIH-103 inhalation solution).

Part C: was an open-label, multi center design study with exploratory objectives to explore the feasibility of patient-led self administration of flecainide. Part C also included an exploratory sub-study to assess the feasibility of implementing a portable cardiac ultrasound (HHE) at screening in an emergent setting.

Upon return to the clinic with a recurrent episode of AF, eligibility was reconfirmed and the subjects self-administered the study treatment and inhalation regimen under medical supervision.

If at 90 minutes after initiation of dosing, no conversion to sinus rhythm (SR) was observed, the Investigator was allowed to offer the subject another appropriate therapy. Discharge was left up to the discretion of the treating physician but no less than 90 min after initiation of dosing. Heart rhythm was confirmed with an Event Recorder during follow up.

An independent Data and Safety Monitoring Board (DSMB) was responsible for monitoring safety during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with recent-onset symptomatic AF at presentation,
2. With a duration at onset of symptoms from 1 hour to 48 hours,
3. And from one of the following categories:

   1. First detected episode of paroxysmal AF
   2. Recurrent episode of paroxysmal AF
   3. Episode post-cardiac ablation for paroxysmal AF

Subjects who:

* are prescribed a pill-in-the-pocket regimen (flecainide or propafenone) for paroxysmal AF, or
* are within 3 months of having undergone ablation of paroxysmal AF, or
* have experienced an episode of new AF but are not currently experiencing an episode of recent-onset paroxysmal AF, or
* are known to have paroxysmal AF (or previously diagnosed with paroxysmal AF) and have one or more previous symptomatic episodes but are not currently experiencing an episode of recent-onset paroxysmal AF may consent to pre-study screening prior to presenting with recent-onset symptomatic AF. These subjects will be eligible to receive study drug only when presenting with symptomatic paroxysmal AF of recent-onset (i.e., ≤ 48 hours), consenting to the full study, and after meeting all eligibility criteria.

Exclusion Criteria:

1. Subject < 18 or > 85 years of age
2. Hemodynamic and/or cardiac instability, with systolic blood pressure < 100 mmHg or > 150 mmHg, and/or ventricular heart rate < 80 bpm or > 150 bpm. For subjects to meet eligibility criteria, at least 2 of the 3 measurements of vital signs during screening (45, 30, and/or 15 minutes prior to dosing) must meet criteria.
3. Current AF episode treated with Class I or Class III antiarrhythmic drugs or electrical cardioversion. Subjects whose current AF episode has been treated with flecainide are eligible if their total cumulative exposure to flecainide (including the study drug to be administered in this study) does not exceed 320 mg within a 24-hour period, per site standard of care.
4. History of acute decompensated heart failure (HF)
5. History within 6 months prior to screening of, or present HF with a left ventricular ejection fraction (LVEF) < 45%, and/or Class II or higher HF as defined by the New York Heart Association (NYHA), and/or medication history suggestive of HF, in the opinion of the Investigator. An echocardiogram with LVEF within 6 months of screening is required to demonstrate eligibility. If no echocardiogram is available, subject must undergo a diagnostic echocardiogram using a portable handheld ultrasound device (handheld echocardiogram; HHE) during screening to confirm eligibility.
6. Evidence of current ongoing myocardial ischemia, such as signs (e.g., significant [e.g., > 2 mm] ST segment elevation or depression on ECG, echocardiographic findings suggestive of acute myocardial infarction), symptoms (e.g., angina pectoris, atypical angina pectoris), and/or being medicated with anti-anginal medication. In addition, subjects with signs of prior myocardial infarction (such as pathological Q waves) who are also taking concomitant medications for angina pectoris should be evaluated for presence of ongoing ischemia.
7. History of myocardial infarction (MI) within 3 months of screening
8. Known uncorrected severe aortic or mitral stenosis
9. Hypertrophic cardiomyopathy with outflow tract obstruction
10. Current diagnosis of persistent AF
11. One or more episodes of atrial flutter within 6 months prior to screening or atrial flutter at presentation
12. History of any of the following heart abnormalities:

    1. Long QT syndrome
    2. Conduction disease (e.g. second- or third- degree heart block, bundle brach block)
    3. Diagnosed with sinus node dysfunction (e.g., sick sinus syndrome) and/or one of the following:

    (i) history of unexplained or cardiovascular syncope, (ii) known bradycardia suggestive of sinus node dysfunction, and/or (iii) prior electrical or pharmacological cardioversion associated with prolonged sinus or ventricular pause (e.g., >3 seconds) and/or slow ventricular rhythm (e.g., <45 bpm) at time of conversion Note: Sinus node dysfunction in AF is more prevalent in subjects >75 years old. d) Brugada Syndrome e) Torsades de pointes (TdP)
13. Any of the following ECG-related features:

    1. QTc interval >480 msec at screening (estimated by the Fridericia's formula)
    2. QRS duration ≥ 120 ms or history of previous documented wide QRS tachycardia
    3. Predominantly (i.e., >30%) paced heart rhythm
    4. Ventricular tachycardia (VT, sustained or non-sustained), or excessive premature ventricular complexes (PVCs, > 20 multifocal PVCs per hour), prior to dosing as per site telemetry. Site telemetry should be equipped with an alarm system for VT and PVCs or be continuously visually observed prior to dosing
14. Severe renal impairment (eGFR < 30 mL/min/1.73 m2) or on dialysis
15. Known abnormal liver function prior to randomization/allocation (including hepatic disease or biochemical evidence of significant liver derangement known prior to randomization/allocation)
16. Uncorrected hypokalemia (defined as serum potassium <3.6 mEq/L) at screening. If serum potassium result is <3.8 mEq/L at screening, therapeutic correction (e.g., potassium supplementation) is strongly encouraged, although reassessing the serum potassium level is not required as long as a value ≥ 3.6 mEq/L is documented at screening.
17. Subjects with established pulmonary disease in need of inhalation medication. Subjects with COPD are excluded. Subjects with mild to moderate asthma that are not experiencing active symptoms at screening and whose asthma is well controlled with steroids and/or as-needed administration of a bronchodilator are eligible for the study.
18. Known hypersensitivity to flecainide acetate or any of its active metabolites
19. Concomitant therapy with systemic drugs that are strong inhibitors of CYP 2D6 (e.g. antidepressants, neuroleptics, ritonavir, some antihistamines) or CYP 2D6 inducers (e.g. phenytoin, phenobarbital, carbamazepine)
20. Treatment with Class I or Class III antiarrhythmic drugs within the last week. Subjects whose current AF episode has been treated with flecainide are eligible if their total cumulative exposure to flecainide (including the study drug to be administered in this study) does not exceed 320 mg within a 24-hour period, per site standard of care.
21. Treatment with amiodarone within the last 12 weeks
22. Subject is deemed unsustainable for the trial by the Investigator (including but not limited to: patients who are considered at high risk for stroke based on screening coagulation panel or medical history (e.g., CHA2DS2-VASc score); patients with congenital heart disease; patients with history of AF refractory to pharmacological or electrical cardioversion; patients whose AF is secondary to electrolyte imbalance, thyroid disease, or other reversible or non-cardiovascular cause; patients with episodes of syncope; patients with any serious or life threatening medical condition; patients with any acute infection). The subject may be deemed unsuitable for the trial by the Investigator if the subject is not able or willing to inhale the study drug.
23. Known drug or alcohol dependence within the past 12 months as judged by the Investigator
24. A body mass index > 40 Kg/m2
25. Legally incompetent to provide informed consent (IC)
26. Previous randomization/allocation in this study or treatment with any other investigational drug within 30 days from screening or 5 half-lives of the drug, whichever is longer
27. Female of childbearing potential

    1. Who are not surgically sterile, or post-menopausal (defined as no menses for 2 years without an alternative cause), or
    2. For whom a negative pregnancy test is unavailable before study entry, or
    3. Who are pregnant or breast feeding at study entry
28. Previous administration of flecainide for an episode of paroxysmal AF or new AF did not result in conversion of AF to SR (i.e., subject is considered a non-responder to flecainide)
29. Cardiac surgery for any of the exclusionary conditions (e.g., valvular disease, hypertrophy, coronary artery disease [CAD], etc.) within the last 6 months prior to screening
30. Respiratory rate of > 22 breaths per minute

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Belardinelli, MD, Study Director — Chief Medical Officer at InCarda Therapeutics
Locations (9):
- Imelda, Bonheiden, Belgium
- Netherlands (8):
  - OLVG, Amsterdam
  - Deventer Ziekenhuis, Deventer
  - Admiraal De Ruyter Ziekenhuis, Goes
  - UMCG, Groningen
  - Spaarne Gasthuis, Haarlem
  - Maastricht University Medical Center, Maastricht
  - Gelre Ziekenhuizen, Zutphen
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruskin JN, Camm AJ, Dufton C, Woite-Silva AC, Tuininga Y, Badings E, De Jong JSSG, Oosterhof T, Aksoy I, Kuijper AFM, Van Gelder IC, van Dijk V, Nuyens D, Schellings D, Lee MY, Kowey PR, Crijns HJGM, Maupas J, Belardinelli L; INSTANT Investigators. Orally Inhaled Flecainide for Conversion of Atrial Fibrillation to Sinus Rhythm: INSTANT Phase 2 Trial. JACC Clin Electrophysiol. 2024 Jun;10(6):1021-1033. doi: 10.1016/j.jacep.2024.02.021. Epub 2024 Apr 10. PMID 38613545
- [Derived] Crijns HJGM, Elvan A, Al-Windy N, Tuininga YS, Badings E, Aksoy I, Van Gelder IC, Madhavapeddi P, Camm AJ, Kowey PR, Ruskin JN, Belardinelli L; INSTANT Investigators*. Open-Label, Multicenter Study of Flecainide Acetate Oral Inhalation Solution for Acute Conversion of Recent-Onset, Symptomatic Atrial Fibrillation to Sinus Rhythm. Circ Arrhythm Electrophysiol. 2022 Mar;15(3):e010204. doi: 10.1161/CIRCEP.121.010204. Epub 2022 Feb 24. PMID 35196871

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A - 30 mg Dose Group: Part A single administration of 30 mg flecainide acetate oral inhalation solution (FlecIH-102) for acute conversion of recent onset of paroxysmal AF to SR
- Part A- 60 mg Dose Group: Part A repeat dose administration of 60 mg flecainide acetate oral inhalation solution (FlecIH-102) for acute conversion of recent onset of paroxysmal AF to SR
- Part A- 90 mg Dose Group: Part A repeat administration of 90 mg flecainide acetate oral inhalation solution (FlecIH-102) for acute conversion of recent onset of paroxysmal AF to SR
- Part A- 120 mg Dose Group Using FlecIH-102: Part A repeat administration of 120 mg flecainide acetate oral inhalation solution (FlecIH-102) for acute conversion of recent onset of paroxysmal AF to SR
- Part A- 120 mg Dose Group Using FlecIH-103: Part A repeat administration of 120 mg flecainide acetate oral inhalation solution (FlecIH-103) for acute conversion of recent onset of paroxysmal AF to SR
- Part B- Dose Confirmation Using 120 mg of FlecIH-103: Part B was designed to confirm the safety and efficacy of the optimal dose and inhalation solution selected in Part A. Patients received 120 mg of FlecIH-103 for acute cardioversion of AF to SR.
- Part C- Cohort Expansion With Exploratory Evaluation of Hand Held Echo: Part C was designed to expand the cohort for medically-led administration of 120 mg of flecainide acetate inhalation solution (FlecIH-103) and to explore the feasibility of patient-led self-administration of flecainide acetate inhalation solution in a hospital setting under medical supervision. The feasibility of implementing a portable cardiac ultrasound (handheld echocardiogram [HHE]) was assessed at screening.
Period: Overall Study
Arm/Group | Part A - 30 mg Dose Group | Part A- 60 mg Dose Group | Part A- 90 mg Dose Group | Part A- 120 mg Dose Group Using FlecIH-102 | Part A- 120 mg Dose Group Using FlecIH-103 | Part B- Dose Confirmation Using 120 mg of FlecIH-103 | Part C- Cohort Expansion With Exploratory Evaluation of Hand Held Echo
Started | 10 | 22 | 21 | 19 | 29 | 26 | 45
Completed | 10 | 22 | 21 | 19 | 29 | 25 | 44
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Spontaneous cardio version | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Part A- Dose Escalation 30 mg FlecIH-102: To evaluate the feasibility of single administration of 30 mg flecainide acetate oral inhalation solution, FlecIH-102 for acute conversion of recent onset of paroxysmal AF to SR.
- Part A- Dose Escalation 60 mg FlecIH-102: To evaluate the feasibility of repeat administration of 60 mg flecainide acetate oral inhalation solution, FlecIH-102 for acute conversion of recent onset of paroxysmal AF to SR.
- Part A- Dose Escalation 90 mg FlecIH-102: To evaluate the feasibility of repeat administration of 90 mg flecainide acetate oral inhalation solution, FlecIH-102 for acute conversion of recent onset of paroxysmal AF to SR.
- Part A- Dose Escalation 120 mg FlecIH-102: To evaluate the feasibility of repeat administration of 120 mg flecainide acetate oral inhalation solution, FlecIH-102 for acute conversion of recent onset of paroxysmal AF to SR.
- Part A- Dose Escalation 120 mg FlecIH-103: To evaluate the feasibility of repeat administration of 120 mg flecainide acetate oral inhalation solution, FlecIH-103 for acute conversion of recent onset of paroxysmal AF to SR.
- Part B- Dose Confirmation: Part B was designed to confirm the safety and efficacy of the optimal dose (120 mg) selected in Part A using FlecIH-103.
- Part C- Cohort Expansion With Exploratory Evaluation of a Hand Held Echo Device: Part C was designed to expand the cohort for medically-led administration of flecainide acetate inhalation solution and to explore the feasibility of patient-led self-administration of flecainide acetate inhalation solution in a hospital setting under medical supervision. Part C also included the evaluation of handheld echo device used at bedside to assess feasibility of its use during screening in an emergent setting.
- Total: Total of all reporting groups
Arm/Group | Part A- Dose Escalation 30 mg FlecIH-102 | Part A- Dose Escalation 60 mg FlecIH-102 | Part A- Dose Escalation 90 mg FlecIH-102 | Part A- Dose Escalation 120 mg FlecIH-102 | Part A- Dose Escalation 120 mg FlecIH-103 | Part B- Dose Confirmation | Part C- Cohort Expansion With Exploratory Evaluation of a Hand Held Echo Device | Total
Number analyzed (Participants) | 10 | 22 | 21 | 19 | 29 | 25 | 44 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 17 | 13 | 17 | 13 | 29 | 108
  >=65 years | 3 | 10 | 4 | 6 | 12 | 12 | 15 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 7 | 11 | 10 | 8 | 16 | 58
  Male | 9 | 17 | 14 | 8 | 19 | 17 | 28 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 21 | 18 | 18 | 26 | 24 | 42 | 157
  Not Reported | 2 | 1 | 3 | 1 | 2 | 0 | 0 | 9
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 27 (3.9) | 26 (3.06) | 27 (3.86) | 28 (5.4) | 26 (3.7) | 27 (3.85) | 27 (4.07) | 27 (3.97)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Conversion of Atrial Fibrillation to Sinus Rhythm
Description: To evaluate the conversion of AF to SR and symptom relief by inhaled flecainide acetate inhalation solution, under two oral inhalation dosing regimens in subjects with recent onset of paroxysmal AF. The subjects will be monitored via ECG and telemetry while in the hospital for 90 minutes.
Time Frame: 90 minutes
Population: Modified Intent to Treat (mITT)
Measure: Number; unit: percentage of participants
Groups:
- Part A- Dose Escalation (30 mg); Part A- Dose Escalation (60 mg); Part A- Dose Escalation (90 mg); Part A- Dose Escalation (120 mg) FlecIH-102; Part A- Dose Escalation (120 mg) FlecIH-103: Part A was designed to evaluate the feasibility of single and repeat administration of escalating doses of flecainide acetate oral inhalation solutions for acute conversion of recent onset of paroxysmal AF to SR.
- Part B- Dose Confirmation: Part B was designed to confirm the safety and efficacy of the optimal dose selected in Part A
- Part C- Cohort Expansion With Exploratory Evaluation of Handheld Echo: Part C was designed to expand the cohort for medically-led administration of flecainide acetate inhalation solution and to explore the feasibility of patient-led self-administration of flecainide acetate inhalation solution in a hospital setting under medical supervision. The feasibility of the use a handheld echo device was assessed during screening in an emergent setting.
Arm/Group | Part A- Dose Escalation (30 mg) | Part A- Dose Escalation (60 mg) | Part A- Dose Escalation (90 mg) | Part A- Dose Escalation (120 mg) FlecIH-102 | Part A- Dose Escalation (120 mg) FlecIH-103 | Part B- Dose Confirmation | Part C- Cohort Expansion With Exploratory Evaluation of Handheld Echo
Number analyzed (Participants) | 10 | 20 | 21 | 17 | 27 | 24 | 43
percentage of participants | 10 | 35 | 33 | 41 | 48 | 50 | 35

2. Secondary Outcome: PK Objectives by Analyzing Blood Samples to Evaluate Peak Plasma Concentration (Cmax)
Description: To explore the population pharmacokinetics (PK) of inhaled flecainide under two oral inhalation dosing regimens in subjects with recent onset paroxysmal AF. Blood samples are collected from each subject for pharmacokinetic analysis.
Time Frame: 90 minutes
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part A 30 mg: Part A 30 mg dose group
- Part A 60 mg: Part A 60 mg dose group
- Part A 90 mg: Part A 90 mg dose group
- Part A 120 mg Using FlecIH-102: Part A 120 mg dose group using FlecIH-102
- Part A 120 mg Using FlecIH-103: Part A 120 mg dose group using FlecIH-103
- Part B Dose Confirmation Using FlecIH-103: To confirm the 120 mg dose using FlecIH-103
- Part C 120 mg Dose Cohort: 120 mg dose cohort using the final formulation, FlecIH-103.
Arm/Group | Part A 30 mg | Part A 60 mg | Part A 90 mg | Part A 120 mg Using FlecIH-102 | Part A 120 mg Using FlecIH-103 | Part B Dose Confirmation Using FlecIH-103 | Part C 120 mg Dose Cohort
Number analyzed (Participants) | 10 | 22 | 21 | 19 | 29 | 25 | 44
ng/mL | 127 (99.5) | 213 (217.3) | 262 (28.7) | 408 (263) | 387 (209.1) | 323.4 (217.8) | 381.5 (236.6)

3. Secondary Outcome: Pharmacodynamics (PD) Objectives by Performing Serial 12-Lead ECG Recordings (Changes in QRS)
Description: To explore the electrocardiographic effects of inhaled flecainide under two oral inhalation dosing regimens in subjects with recent onset of paroxysmal AF. Serial 12-Lead ECG measurements are extracted from the Holter recording in triplicate before, after the allocated inhalation regimen and at the time of conversion to sinus rhythm for pharmacodynamic analysis.
Time Frame: 90 minutes
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Part A 30 mg: Part A 30 mg dose group using the FlecIH-102 inhalation solution
- Part A 60 mg: Part A 60 mg dose group using the FlecIH-102 inhalation solution
- Part A 90 mg: Part A 90 mg dose group using the FlecIH-102 inhalation solution
- Part A 120 mg Using FlecIH-102: Part A 120 mg dose group using the FlecIH-102 inhalation solution
- Part B 120 mg Using FlecIH-103: Part B 120 mg dose group using FlecIH-103 inhalation solution
- 120 mg Dose Group Part C: The analyses of the 120 mg dose cohort using the final formulation, FlecIH-103.
Arm/Group | Part A 30 mg | Part A 60 mg | Part A 90 mg | Part A 120 mg Using FlecIH-102 | Part A 120 mg Using FlecIH-103 | Part B 120 mg Using FlecIH-103 | 120 mg Dose Group Part C
Number analyzed (Participants) | 10 | 22 | 21 | 19 | 29 | 25 | 44
msec | 4.3 (13.6) | 2.6 (4.9) | 2.9 (3.1) | 7.9 (8.1) | 6.6 (4.2) | 7.0 (9.3) | 4.5 (4.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through Day 5.
Description: The study collected adverse events of special interest which included events related to the device, pregnancy, AEs known to other formulations of flecainide, hypotension (BP < 90/60 mmHg ), ventricular tachycardia (≥ 3 beats), Bradycardia (rate < 50 bpm for ≥ 1 minute), Sinus pauses post conversion of AF to SR: an ECG-derived pause > 3 seconds, Atrial flutter with 1:1 conduction with fast ventricular response (ventricular heart rate ≥ 200 bpm)
Groups:
- Part A 30 mg Dose Using FlecIH-102: 30 mg dose using FlecIH-102 for acute cardioversion of AF to SR
- Part A 60 mg Dose Using FlecIH-102: 60 mg dose using FlecIH-102 for acute cardioversion of AF to SR
- Part A 90 mg Dose Using FlecIH-102: 90 mg dose using FlecIH-102 for acute cardioversion of AF to SR
- Part A 120 mg Dose Using FlecIH-102: 120 mg dose using FlecIH-102 for acute cardioversion of AF to SR
- Part A 120 mg Dose Using FlecIH-103: 120 mg dose using FlecIH-103 for acute cardioversion of AF to SR
- Part B 120 mg Dose Using FlecIH-103: Dose confirmation cohort for 120 mg dose group using the final formulation of study drug, FlecIH-103.
- Part C 120 mg Dose Using FlecIH-103: Dose expansion cohort for 120 mg dose using the final formulation of study drug, FlecIH-103.
Arm/Group | Part A 30 mg Dose Using FlecIH-102 | Part A 60 mg Dose Using FlecIH-102 | Part A 90 mg Dose Using FlecIH-102 | Part A 120 mg Dose Using FlecIH-102 | Part A 120 mg Dose Using FlecIH-103 | Part B 120 mg Dose Using FlecIH-103 | Part C 120 mg Dose Using FlecIH-103
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/22 | 0/21 | 0/19 | 0/29 | 0/25 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/10 | 3/22 | 1/21 | 1/19 | 2/29 | 2/25 | 0/44
Other Adverse Events (participants affected / at risk) | 9/10 | 16/22 | 17/21 | 16/19 | 25/29 | 17/25 | 23/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A 30 mg Dose Using FlecIH-102 (N=10) | Part A 60 mg Dose Using FlecIH-102 (N=22) | Part A 90 mg Dose Using FlecIH-102 (N=21) | Part A 120 mg Dose Using FlecIH-102 (N=19) | Part A 120 mg Dose Using FlecIH-103 (N=29) | Part B 120 mg Dose Using FlecIH-103 (N=25) | Part C 120 mg Dose Using FlecIH-103 (N=44)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter with 1:1 AV conduction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfuntion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (hospitalization for recurrence of AF) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus arrest/Ventricular systole (asystolic pause) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A 30 mg Dose Using FlecIH-102 (N=10) | Part A 60 mg Dose Using FlecIH-102 (N=22) | Part A 90 mg Dose Using FlecIH-102 (N=21) | Part A 120 mg Dose Using FlecIH-102 (N=19) | Part A 120 mg Dose Using FlecIH-103 (N=29) | Part B 120 mg Dose Using FlecIH-103 (N=25) | Part C 120 mg Dose Using FlecIH-103 (N=44)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3)
Salivary Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (9) | 11 (11) | 13 (13) | 12 (12) | 11 (11) | 15 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (4) | 4 (4) | 4 (4) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Condition aggravated (General disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SV extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SV tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular Systole (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT03539302/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT03539302/SAP_002.pdf